CLINICAL TRIAL: NCT01594879
Title: Treatment With Medroxyprogesterone Acetate(MPA) Plus Levonorgestrel-releasing Intrauterine System(LNG-IUS) in Young Women With Early Stage Endometrial Cancer: Multicenter Study: Korean Gynecologic Oncology Group Study (KGOG2009)
Brief Title: Treatment With Medroxyprogesterone Acetate Plus LNG-IUS in Young Women With Early Stage Endometrial Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korean Gynecologic Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KGOG2009
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer; LNG-IUS; oral MPA
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endometrial cancer, LNG-IUS with MPA (Experimental)
  Interventions: Device: MIrena(LNG-IUS), oral MPA

INTERVENTIONS:
Device: MIrena(LNG-IUS), oral MPA — 1. General Name/Brand name: Mirena - SCHERING Active ingredient: levonorgestrel 52mg Description: Mirena is a hormone-releasing T-shaped intrauterine system. A removal thread is attached to a loop at the end of the vertical stem of the T-body.
  2. General Name/Brand name:Farlutal tab. 500mg/ Pfizer Active ingredient: Medroxyprogesterone Acetate
  Other Names: Mirena; Farlutal

SUMMARY:
A prospective multicenter trial has been started in Korea to investigate the treatment efficacy of Levonorgestrel-releasing intrauterine system (LNG-IUS) plus Medroxyprogesterone Acetate(MPA) in Young Women with Early Stage Endometrial Cancer.

The standard treatment for endometrial cancer is total hysterectomy and bilateral salpingo-oophorectomy, peritoneal cytology, and lymph node dissection. However, young patients who desire to preserve their potential for fertility may find this standard treatment difficult to accept. Therefore, the conservative treatment for these patients has remained a challenge. A number of studies have reported the effectiveness of hormonal therapy using systemic progestin in women clinically diagnosed with early endometrial adenocarcinoma at stage IA, grade 1, who want to maintain reproductive potential. In addition, several recent studies reported the use of LNG-IUS to treat patients at a high risk of perioperative complications who cannot tolerate systemic progesterone because of its adverse effects. Nevertheless, there has been no prospective multicenter trial that investigated the effectiveness of treatment with systemic progesterone in combination with intrauterine progesterone in young women with endometrial cancer.

Therefore, the investigators conducted a prospective trial of the treatment of the presumably early-stage grade 1 endometrial cancer in young women who desire to preserve fertility by using oral MPA in combination with LNG-IUS.

Young patients with histologically confirmed grade 1 endometrioid adenocarcinoma that is presumably confined to the endometrium, who desired to preserve fertility potential go through LNG-IUS insertion and are administered MPA at a dosage of 500 mg/d concurrently. Follow-up and treatment response assessment were implemented at a 3-month interval with office endometrial aspiration biopsy with LNG-IUS in place and dilatation and curettage after removal of LNG-IUS.

The primary endpoint is response rate. Secondary endpoint is to estimate the consistency of the results between office endometrial aspiration biopsy and dilatation and curettage (D&C) procedure.

DETAILED DESCRIPTION:
PURPOSE: This prospective study aims to analyze the treatment efficacy of LNG-IUS plus MPA in Young Women with Early Stage Endometrial Cancer and to analyze the diagnostic accuracy of office endometrial aspiration biopsy with LNG-IUS in place compared with dilatation and curettage after removal of LNG-IUS.

ENDPOINTS: The primary endpoints of this study is response rate. Secondary endpoint is to estimate the consistency of the results between office endometrial aspiration biopsy and dilatation and curettage (D&C) procedure.

STUDY SETTING AND PROTOCOL REVIEW: This study is a single arm, prospective multi-institutional study. Its protocol was approved by the Institutional Review Board of each clinical trial institution.

PLANNED CLINICAL TRIAL PERIOD: Patient Selection and Enrollment: 24 month after IRB approval of clinical trial Institution.

TREATMENT METHODS: Patients with histologically confirmed grade 1 endometrioid adenocarcinoma that is presumably confined to the endometrium went through LNG-IUS insertion and were administered MPA at a dosage of 500 mg/day concurrently. Follow-up and treatment response assessment were implemented at a 3-month interval with transvaginal ultrasonography, endometrial aspiration biopsy with LNG-IUS in place and D&C after removal of LNG-IUS. The biopsy findings are compared.

INVESTIGATIONAL PRODUCT

1. General Name/Brand name: Mirena - SCHERING

   Active ingredient: levonorgestrel 52mg

   Description: Mirena is a hormone-releasing T-shaped intrauterine system. A removal thread is attached to a loop at the end of the vertical stem of the T-body.
2. General Name/Brand name:Farlutal tab. 500mg/ Pfizer

Active ingredient: Medroxyprogesterone Acetate

PLANNED NUMBER OF SUBJECT 39 patients with biopsy proven grade 1 endometrioid adenocarcinoma that is presumably confined to the endometrium.

STATISTICAL CONSIDERATIONS The primary objective of this study is to estimate the treatment efficacy of the oral MPA in combination with LNG-IUS in early stage endometrial cancer in terms of their response rate. The sample size needed for this estimation would be 39 patients after considering 10% of follow-up loss. The Secondary objective is to estimate the consistency of the office endometrial aspiration biopsy and D&C. Kappa statistics will be used

ELIGIBILITY:
Inclusion Criteria:

1. Patients younger than 40 years
2. Patients who are histological confirmed as endometrial adenocarcinoma grade I that is presumably confined to the endometrium based on the MRI evaluation
3. Patients who desire to preserve fertility potential
4. Patients signed the written informed consent voluntarily

Exclusion Criteria:

1. Patients who have severe underlying disease or complication
2. Under treatment of metastatic cancer from other organs or less than 5 years after previous cancer therapy
3. Acute liver disease or kidney disease
4. Thrombosis or phlebothrombosis requiring treatment, Hyperlipidemia, Smoker

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
response rate | 24months after LNG-IUS insertion with taking oral MPA
  Young patients with histologically confirmed grade 1 endometrioid adenocarcinoma that is presumably confined to the endometrium, who desired to preserve fertility potential go through LNG-IUS insertion and are administered MPA at a dosage of 500 mg/d concurrently.
  Follow-up and treatment response assessment were implemented at a 3-month interval with office endometrial aspiration biopsy with LNG-IUS in place and dilatation and curettage after removal of LNG-IUS.

SECONDARY OUTCOMES:
consistency of the results between office endometrial aspiration biopsy and dilatation and curettage (D&C) procedure. | every 3 month after LNG-IUS insertion with taking oral MPA
  consistency of the results between office endometrial aspiration biopsy and dilatation and curettage (D&C) procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Seok Ju Seong, MD, Principal Investigator — Gangnam CHA medical center
Locations (1):
- Gangnam CHA medical center, Seoul, Gamnamgu, South Korea

REFERENCES:
- [Derived] Kim MK, Seong SJ, Kang SB, Bae DS, Kim JW, Nam JH, Lim MC, Lee TS, Kim S, Paek J. Six months response rate of combined oral medroxyprogesterone/levonorgestrel-intrauterine system for early-stage endometrial cancer in young women: a Korean Gynecologic-Oncology Group Study. J Gynecol Oncol. 2019 Mar;30(2):e47. doi: 10.3802/jgo.2019.30.e47. Epub 2019 Jan 7. PMID 30740964